CLINICAL TRIAL: NCT02700243
Title: Pilot RCT Study Using a Fitbit Device to Improve Exercise Tolerance in 80 Patients With Cystic Fibrosis
Brief Title: Increase Tolerance for Exercise and Raise Activity Through Connectedness Trial
Acronym: INTERACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Uluer, Director, Adult Cystic Fibrosis Program, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00012871
Record Dates: First submitted 2016-02-21; First posted 2016-03-07 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Exercise; Fitbit
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fitbit (Experimental): Participants receive a Fitbit and are followed over the course of one year, completing surveys and exercise tests.
  Interventions: Behavioral: Fitbit
- Usual Care (No Intervention): Participants receive usual care over the course of one year and are offered a Fitbit in the second year. Followed to assess use of Fitbit and health outcomes.

INTERVENTIONS:
Behavioral: Fitbit — Participants receive a Fitbit and are followed over the course of one year to determine use and health outcomes.
  Arms: Fitbit

SUMMARY:
In this research study the investigators want to learn more about whether using a fitness tracker and accelerometer helps patients with cystic fibrosis exercise more regularly, and in turn whether it increases exercise tolerance over the period of one year.

DETAILED DESCRIPTION:
The aim of this study is to evaluate whether the use of a Fitbit device and an exercise prescription is associated with increased daily activity and in turn increased exercise tolerance in young adult patients with cystic fibrosis (CF). The investigators hypothesize that use of the Fitbit and an exercise prescription will be associated with increased exercise tolerance compared to standard counseling and an exercise prescription alone.

For patients with CF, young adulthood and adolescence is a significant time of vulnerability. In addition to normal behavioral challenges of adolescence and young adulthood (seeking independence/autonomy while also choosing rebellion), those with CF are often dealing with significant disease progression. Therefore, working in new innovative ways to improve adherence to regimens that improve lung function such as exercise are needed to continue to support patients during this vulnerable time.

Studies of patients with cystic fibrosis have shown that regular exercise training can decrease rate of lung function decline, potentially improve lung function, and improve aerobic capacity. However, many patients do not include regular exercise in their daily routine. Successful strategies to improve adherence include providing patient specific guidelines for an appropriate exercise program, supporting participation and providing positive feedback. Overall, exercise is a crucial diagnostic and therapeutic modality for patients with Cystic Fibrosis, although awareness somewhat limited. The adult CF program at Boston Children's and Brigham & Women's Hospital established an inpatient and outpatient exercise program as part of a quality improvement effort. Patients are prescribed an individualized exercise program or exercise prescription based on their assessment during a sub-maximal effort. This program has been successful but given the rigors of daily life (e.g. school, work, family obligations), adherence is a concern with resources limiting more rigorous feedback to maintain this essential life activity.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of Cystic Fibrosis
2. Age 18 and over
3. Must be able to complete at least level 1 of the baseline exercise fitness test
4. Must not have required IV antibiotics for a CF exacerbation within 30 days of starting the program

Exclusion Criteria:

1. Pregnancy at enrollment
2. A history of CF exacerbation requiring IV antibiotics within last month
3. Use of a fitness tracker or similar product within 6 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Graded exercise test (Submaximal GXT) | Two years (Enrollment, 6 months, 12 months, 24 months)
  Change is submaximal GXT will be assessed for all participants

SECONDARY OUTCOMES:
Fitbit activity data | Two years
HAES (Habitual Activity Estimation Scale) | Two years
Relative change from baseline in ppFEV1 | Two years
  Forced Expiratory Volume in one second (FEV1) from before study (Baseline) to each data collection timepoint, and from one data collection timepoint to the next.
Relative change from baseline in ppFVC | Two years
  Forced Vital Capacity in one second (FVC) from before study (Baseline) to each data collection timepoint, and from one data collection timepoint to the next.
Relative change from baseline in ppFEF25-75 | Two years
  Forced Expiratory Flow in one second (FEF25-75) from before study (Baseline) to each data collection timepoint, and from one data collection timepoint to the next.
Incidence of exacerbations requiring IV antibiotics | Two years
BMI | Two years
CFQ-R (Survey on Quality of Life in Cystic Fibrosis) | Two years
Overall qualitative assessment of participant satisfaction with the Fitbit | Two years (6 Month Time Point)
  Qualitative data obtained by open-ended interview
Overall qualitative assessment of participant's potential barriers to Fitbit use | Two years (6 Month Time Point)
  Qualitative data obtained by open-ended interview
Overall qualitative assessment of the participant's use of the social media associated with the device | Two years (6 Month Time Point)
  Qualitative data obtained by open-ended interview
PHQ9 | Two years (Enrollment, 6 months, 12 months, 18 months, 24 months)
  Depression scale scored 0-27, with a score of 0-4 indicating minimal risk for depression/anxiety, a score of 5-9 indicating mild risk for depression/anxiety, a score of 10-14 indicating moderate risk for depression/anxiety, and a score if 15-27 indicating severe risk for depression/anxiety.
GAD-7 | Two years (Enrollment, 6 months, 12 months, 18 months, 24 months)
  Depression scale scored 0-21, with a score of 0-4 indicating minimal risk for depression/anxiety, a score of 5-9 indicating mild risk for depression/anxiety, a score of 10-14 indicating moderate risk for depression/anxiety, and a score if 15-21 indicating severe risk for depression/anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Uluer, DO, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: Yes
Participants will receive their graded exercise test scores as part of their clinical care and will be able to see their individual data relating to Fitbit on their own device.